CLINICAL TRIAL: NCT00300326
Title: An Investigation of Total Knee Arthroplasty Kinematics on Patient Performance - The Zimmer Legacy® LPS Flex Knee System
Brief Title: Computer-assisted Total Knee Arthroplasty (TKA) With Zimmer LPS Flex Knee System
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: problems with planned computer
Sponsor: Queen's University (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Dr. John Rudan, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURG-130-04
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2009-04

CONDITIONS: Knee Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Using the same knee implant with a conventional surgical technique.
- 2 (Active Comparator): Using the same knee implant using a computer-assist surgery group is the comparator
  Interventions: Procedure: Computer assist

INTERVENTIONS:
Procedure: Computer assist — same implant using a computer-assisted surgical technique.
  Arms: 2

SUMMARY:
To determine clinical outcomes and biomechanical gait performance of patients who receive the Zimmer Legacy® LPS Flex Knee system using a computer-assisted surgical technique. This study will provide evidence as to whether there are differences between the two surgical procedures with respect to complications such as infection and dislocations, rate and level of functional recovery, blood loss, operating time, degree of radiographic correction and quality and duration of post-operative pain and stiffness.

DETAILED DESCRIPTION:
The objective of this study is to determine the clinical outcomes and biomechanical gait performance of patients who receive the Zimmer Legacy® LPS Flex Knee system using a computer-assisted surgical technique. Pre and post-operative clinical and gait variables will be compared within the computer-assisted group. These same comparisons will also be made between the computer-assisted surgical group and a conventional surgical group who receive the same knee implant. This study will further provide evidence as to whether there are differences between the two surgical procedures with respect to complications such as infection and dislocations, rate and level of functional recovery, blood loss, operating time, degree of radiographic correction and quality and duration of post-operative pain and stiffness.

ELIGIBILITY:
Inclusion Criteria:

* age 50-80

  * undergoing primary total knee arthroplasty
  * femoral tibial varus < 7 degrees
  * no previous joint infections
  * anteriorcruciate ligament intact
  * clinically significant patellofemoral or osteoarthritic degeneration

Exclusion Criteria:

* active articular infections
* significant concurrent ipsilateral hip osteoarthritis
* chronic pain syndrome requiring medications for control
* history of chemical addiction
* significant spinal stenosis, chronic back pain, sciatica
* patients who are unlikely to comply with, participate in or return for follow-up visits as described in the protocol
* osteomyelitis, septicemia or other infections that may spread to other areas of the body
* highly communicable diseases, immuno-compromising conditions and/or that may limit follow-up (eg. AIDS, active tuberculosis, venereal disease, active hepatitis, neoplastic disease)
* diabetic neuropathy
* skeletal immaturity
* decreased mental comprehension and literacy
* pregnancy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-01; Primary Completion 2011-04 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Gait kinetic and kinematic parameters at the knee (knee forces, moments and angles) | pre-op and 1 year

SECONDARY OUTCOMES:
knee pain, stiffness and function | preop- 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Rudan, MD, Principal Investigator — Queen's University